CLINICAL TRIAL: NCT01121354
Title: A Phase I Multiple-Dose Two-Arm Study to Evaluate the PK and Safety of Cefazolin 2g for Inj. USP and Dextrose Inj. USP in the DUPLEX® Drug Delivery System and Cefazolin for Inj. 1.5g in Daily Doses of 6g in Healthy Adult Subjects
Brief Title: Pharmacokinetics and Safety of Cefazolin 2g in DUPLEX
Acronym: 2 Cef
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: B. Braun Medical Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HC-G-H-0906
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Infection
Keywords: Cefazolin; Caphalosporin; antibiotic; gram positive; Infection control
MeSH Terms: conditions — Infections | interventions — Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cefazolin 2g (Test) (Experimental)
  Interventions: Drug: Cefazolin 2g for Injection USP and Dextrose Injection USP
- Cefazolin 1.5g (Control) (Active Comparator)
  Interventions: Drug: Cefazolin 1.5g

INTERVENTIONS:
Drug: Cefazolin 2g for Injection USP and Dextrose Injection USP — Cefazolin 2g for Injection USP and Dextrose Injection USP in the DUPLEX® Drug Delivery System. Administration will occur three times per day (t.i.d.) over an eleven (11) day period, with nine (9) days of repeated dosing.
  Other Names: Cefazolin 2g in DUPLEX (50ml)
  Arms: Cefazolin 2g (Test)
Drug: Cefazolin 1.5g — Cefazolin 1.5g for Injection USP and Dextrose Injection USP in a pharmacy-prepared container. Administration will occur four times per day (q.i.d.) over an eleven (11) day period, with nine (9) days of repeated dosing.
  Other Names: Cefazolin 1.5g (50ml)
  Arms: Cefazolin 1.5g (Control)

SUMMARY:
The purpose of this study is to demonstrate the safety and pharmacokinetics of Cefazolin 2g for Injection USP and Dextrose Injection USP in the DUPLEX® Drug Delivery System to Cefazolin 1.5g for Injection USP and Dextrose Injection USP in daily doses of 6g in healthy adult subjects for 11 days of administration.

DETAILED DESCRIPTION:
B. Braun Medical Inc. intends to conduct human PK studies and obtain marketing approval for Cefazolin 2g in the United States with identical indications of those already approved for the 1g strength. A pharmacokinetic study will be conducted with the Cefazolin 2g product manufactured by B. Braun Medical Inc. Cefazolin 1.5g dose will be prepared using 10g Cefazolin pharmacy bulk with 5% Dextrose. The clinical study proposed in this protocol is designed to evaluate the pharmacokinetic characteristics of 2g and 1.5g Cefazolin in Dextrose in healthy subjects at the maximum recommended infusion dose of 6g per day per FDA's recommendation.

The study is designed to simulate clinical practice and overall experience with cephalosporin administration. Cefazolin may be reconstituted with dextrose (or a number of other diluents as recommended in the innovator's package insert) in order to achieve an osmolality appropriate for intravenous infusion.

According to B. Braun's approved package insert for Cefazolin 1g, the maximum dose of 1.5g Cefazolin for Injection USP and Dextrose Injection USP is 1.5 grams every 6 hours for severe, life-threatening infections. In rare instances, doses of up to 12 grams of Cefazolin per day have been used. Lower doses are stated in the B. Braun package insert.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, male and female
* Age: 18 - 70 years (inclusive) at the time of screening.
* Females of non-child bearing potential (surgically sterile [hysterectomy or bilateral tubal ligation] or post-menopausal >= 1 year with follicle stimulating hormone [FSH] > 40 U/L).
* Healthy, determined by pre-study medical evaluation (medical history, physical examination, vital signs, electrocardiogram, and clinical laboratory evaluations).
* Subject voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB)-approved informed consent and the Health Insurance Portability and Accountability Act (HIPAA) Authorization prior to performing any of the screening procedures.

Exclusion Criteria:

* Known allergy or hypersensitivity to beta-lactam/cephalosporin antibiotics, corn products or any of the other ingredients of the Investigational Products
* Subjects with impaired renal function based on the Cockcroft-Gault formula using actual body weight, i.e. estimated creatinine clearance <= 80 mL/min (performed at Screening only)
* Body Mass Index (BMI) < 20.0 or > 30.0 kg/m^2
* Body Weight < 50.0 kg
* White Blood Count (WBC) < 3.5 x10^3/uL or > ULN
* absolute neutrophil count (ANC) < 1.5 x10^3/uL or > ULN
* Alarine aminotransferase and aspartate aminotransferase > upper limit of normal
* Other laboratory tests that are outside the normal limits, considered by the investigator, to be clinically significant.
* Use of any medication on a chronic basis.
* Takes any medication which interferes with the study drug or study procedures including aminoglycosides, anticoagulants, and probenecids.
* Use of over the counter (OTC) medications (including vitamins), prescription medications, or herbal remedies from 14 days prior to Day -1 until end of study. By exception, acetaminophen <= 1 gram per day is permitted.
* Tobacco use during the last 2 months prior to enrollment.
* Positive screening test for Hepatitis B surface antigen, Hepatitis C antibody, or human immunodeficiency virus (HIV) antibody.
* Positive urine drug test (cocaine, amphetamines, barbiturates, opiates, benzodiazepines, cannabinoids, etc.) at Screening or Day -1
* Positive blood test for ethanol at screening or Day -1.
* At screening, the subject has a clinically relevant ECG change, as assessed by the PI or designee.
* Concurrent acute or chronic infections (e.g. viral infections, except chronic recurrent herpes infections)
* History of or ongoing alcohol abuse or drug abuse (within last 2 years).
* Received an Investigational drug or device within 30 days of first dose of study drug
* Clinically relevant medical conditions which are likely to interfere with the evaluation of the trial drug, e.g. COPD, metabolic disorders (such as clinical and sub-clinical diabetes mellitus), history of malignant diseases (within last 5 years), autoimmune diseases, and cardiovascular disease
* Any planned medical intervention or personal event that might interfere with the ability to comply with the study requirements
* Any condition that, in the opinion of the principal investigator, would compromise the safety of the patient or the quality of the data
* Unable or unwilling to adhere to the study-specified procedures and restrictions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of an intravenous infusion of Cefazolin 2g in healthy adult subjects at an infusion rate of 50 ml over 15 minutes, and Cefazolin 1.5g in a similar population of healthy adult subjects | PK is evaluated on Days 1 and 11 of infusion therapy
  The primary objective is to evaluate the pharmacokinetics of an intravenous infusion of Cefazolin 2g for injection USP and Dextrose injection USP in healthy adult subjects at an infusion rate of 50 ml over 15 minutes, and Cefazolin 1.5g for injection USP and Dextrose injection USP in a similar population of healthy adult subjects.

SECONDARY OUTCOMES:
To evaluate the safety of cefazolin 2g injection in total daily doses of 6g over 11 days of administration in healthy volunteers | Varies, over 11 days of infusion therapy
  * Hematology(CBC): Hb, Hct, RBC count, RBC indices, RBC morphology, platelet count, WBC count, and differential WBC
  * Clinical Chemistry: Sodium, potassium, chloride, Co2, glucose, ALT, AST, alkaline phosphatase, serum albumin, total bilirubin, blood urea nitrogen, and creatinine
  * Urinalysis: specific gravity, protein, blood, nitrates, leukocyte esterase, glucose, ketone, appearance, pH
  * Urine drug and blood alcohol tests
  * C. difficile
  * ECG
  * Vital signs: temperature, blood pressure, heart rate, and respiratory rate
  * Adverse Events
  * Physical exams

CONTACTS AND LOCATIONS:
Overall Officials: Azra Hussaini, MD, Principal Investigator — Parexel
Locations (1):
- PAREXEL Early Phase Clinical Unit, Baltimore, Maryland, United States

REFERENCES:
- [Background] Abraxis Pharmaceutical Products, Package Insert, Cefazolin for Injection, USP.45858E, July 2006, Schaumburg, IL 60173 (USA).
- [Background] Apotex Corp., Package Insert, Cefazolin for Injection, USP, Pharmacy Bulk Pack. 948025398, December 2005, Weston, FL 33326 (USA).
- [Background] APP Pharmaceuticals, LLC. Package Insert, Cefazolin for Injection, USP. 451180, July 2008, Schaumburg, IL 60173 (USA).
- [Background] Hospira, Inc. Package Insert, Cefazolin for Injection, USP, Pharmacy Bulk Pack. EN-1961/948025777, December 2008, Lake Forest, IL 60045 (USA).
- [Background] B. Braun Medical inc., Package Insert, Cefazolin for Injection USP and Dextrose Injection USP in DUPLEX Container, 1g, Apr 2008, Allentown, PA 18109 (USA).
- [Background] Vella-Brincat JW, Begg EJ, Kirkpatrick CM, Zhang M, Chambers ST, Gallagher K. Protein binding of cefazolin is saturable in vivo both between and within patients. Br J Clin Pharmacol. 2007 Jun;63(6):753-7. doi: 10.1111/j.1365-2125.2006.02827.x. Epub 2007 Jan 12. PMID 17223858